CLINICAL TRIAL: NCT01425736
Title: Phase 2 Study of Nimotuzumab in Combination With TPF for Head and Neck Squamous Cell Carcinoma
Brief Title: Nimotuzumab in Combination With TPF(Cisplatin ,Fluorouracil and Docetaxel) for Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wei Guo (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor-Investigator, Wei Guo, Guo Wei, Shanghai 9th People's Hospital., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-IST-SCCHN-008
Record Dates: First submitted 2011-08-19; First posted 2011-08-30 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Nimotuzumab; Chemotherapy; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy; Docetaxel; Cisplatin; Fluorouracil; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Placebo Comparator): Chemotherapy
  :Docetaxel(75mg/m²,1 time/21d, 6times);Cisplatin(75mg/m²,1 time/21d, 6 times);Fluorouracil(750mg/m²/d,5times/21d, 30times)
  Interventions: Drug: Chemotherapy
- Nimotuzumab and Chemotherapy (Experimental): Nimotuzumab treatment:(200mg/w,18weeks );
  Chemotherapy treatment: Docetaxel(75mg/m²,1 time/21d, 6times，);Cisplatin(75mg/m²,1 time/21d, 6 times);Fluorouracil(750mg/m²/d,5times/21d, 30times),Nimotuzumab treatment:(200mg/w,18weeks ).
  Interventions: Drug: Nimotuzumab and Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy :Docetaxel(75mg/m²,1 time/21d, 6times);Cisplatin(75mg/m²,1 time/21d, 6 times);Fluorouracil(750mg/m²/d,5times/21d, 30times)
  Other Names: Docetaxel; Cisplatin; Fluorouracil
  Arms: Chemotherapy
Drug: Nimotuzumab and Chemotherapy — Nimotuzumab treatment:(200mg/w,18weeks );
  Chemotherapy treatment:(Docetaxel(75mg/m²,1 time/21d, 6times);Cisplatin(75mg/m²,1 time/21d, 6 times);Fluorouracil(750mg/m²/d,5times/21d, 30times)Nimotuzumab treatment:(200mg/w,18weeks );
  Other Names: Docetaxel; Cisplatin; Fluorouracil; Nimotuzumab
  Arms: Nimotuzumab and Chemotherapy

SUMMARY:
Nimotuzumab (hR3) is an humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). In phase II clinical trials a combination of Nimotuzumab with chemotherapy or radiation therapy achieved satisfactory therapeutic outcomes in patients with advanced squamous cell carcinoma of head and neck, or glioblastoma. We therefore postulated that Nimotuzumab in combination with conventional definitive chemotherapy might improve the rate of disease control (RDC), progression-free survival (PFS),and overall survival in patients with recurrent and/or metastatic SCCHN , which is a poor-prognosis patient population for whom there is currently no standard treatment approach, we designed this trial to test this hypothesis.

DETAILED DESCRIPTION:
Eligible patients were randomly assigned by using permutated blocks designed11 for each site to receive either Nimotuzumab combined with docetaxel-cisplatin-fluorouracil regimen (Arm A) or docetaxel-cisplatin-fluorouracil alone regimen (Arm B). Combination arm chemotherapy was as conducted as follows. Since day 1, Nimotuzumab (200 mg, given as a 2-hour intravenous infusion before chemotherapy, Biotech Pharmaceutical Inc., Beijing, China) was administrated 1 h before chemotherapy once a week for two successive courses, followed by docetaxel (at a dose of 75 mg per square meter of body-surface area) was administered as a 1-hour intravenous infusion, followed by intravenous cisplatin (75 mg per square meter), administered during a period of 0.5 to 3 hours. After completion of the cisplatin infusion, fluorouracil (1000 mg per square meter per day) was administered as a continuous 24-hour infusion for 4 days. Patients in arm A received docetaxel-cisplatin-fluorouracil only.One treatment cycle comprised a period of 3 weeks (21 days). Patients received six cycles in both treatment arms, unless disease progression or unacceptable toxicity was observed. Patients in the experimental group who had at least stable disease could choose to continue maintenance Nimotuzumab every week until disease progression, intolerable toxicity, or study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntary and signed informed consent form
* Age 18-75，both genders.
* Had histologically or cytologically confirmed recurrent or metastatic squamous cell carcinoma of the head and neck
* At least one lesions can be measured,Conventional measurements ≥2cm, computed tomography(CT) examination ≥1cm .
* Eastern Cooperative Oncology Group(ECOG) Performance Scale 0-2.
* Life expectancy of more than 3 months.
* Use of an effective contraceptive method for women when there is a risk of pregnancy during the study.
* Haemoglobin≥90g/L ,White blood cell(WBC) ≥3×10^9/L
* Hepatic function:ALAT、ASAT< 2.5 x ULN, TBIL< 1.5 x ULN
* Renal function: Creatinine < 1.5 x ULN

Exclusion Criteria:

* Received other anti EGFR monoclonal antibody treatment
* Participation in other interventional clinical trials within 1 month
* Previous received other drug or operative treatment within 6 month
* Pregnant or breast-feeding women
* History of serious allergic or allergy
* Patients with the history of Serious lung or head disease
* Other malignant tumor
* not primary tumor(except for primary tumor therapy>3months)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Rate of Disease Control (RDC) | 4years

SECONDARY OUTCOMES:
toxicity, progression-free survival (PFS), and overall survival (OS). | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, MD, PhD, DDS, Study Chair — Dept. of Oral and Maxillofacial Surgery,9th People's Hospital, School of Stomatology,Shanghai Jiaotong University
Locations (5):
- China (5):
  - First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Institute of Stomatology of Nanjing Medical University, Nanjing, Jiangsu
  - Wuxi People's Hospital; Nanjing Medical University, Wuxi, Jiangsu
  - Xuzhou Central Hospital of Xuzhou city,Dongnan University, Xuzhou, Jiangsu
  - 9th People's Hospital, School of Stomatology,Shanghai Jiaotong University, Shanghai, Shanghai Municipality